CLINICAL TRIAL: NCT01850563
Title: A Proof-of-principle Study of Hyperbaric Oxygen as a Radiosensitizer Prior to Stereotactic Radiosurgery for Brain Metastases
Brief Title: A Proof-of-principle Study of HBO-SRS for Brain Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Alan Hartford, Staff Physician, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D12129
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Results first posted 2021-07-29 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Brain Metastases
Keywords: Demonstrate coordination of HBO with SRS treatments is feasible.; Demonstrate outcomes for patients treated with combination of HBO and SRS are non-inferior .
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- HBO feasibility (Other)
  Interventions: Device: Hyperbaric oxygen given at 2.4 ATA for 30 minutes immediately prior to SRS - HBOT for 30 minutes - SRS without prior HBO

INTERVENTIONS:
Device: Hyperbaric oxygen given at 2.4 ATA for 30 minutes immediately prior to SRS - HBOT for 30 minutes - SRS without prior HBO

SUMMARY:
Patients with brain metastases who are candidates for treatment with stereotactic radiosurgery (SRS) are potential study participants. SRS delivers high-energy, precisely-focused radiation to each brain metastasis to shrink the tumor, and is the standard-of-care for patients with these tumors. Oxygen enhances the damaging effects of radiation on tumor cells. Hyperbaric oxygen (HBO) therapy increases oxygen levels in all kinds of tissues, including tumors. The purpose of this trial is to study whether it is feasible to treat patients with HBO just prior to receiving SRS, given the timing constraints of treating sequentially with HBO and then SRS. Patients will undergo HBO treatment followed by the placement of a Gill-Thomas-Cosman head frame then transported ,via stretcher, to receive SRS. The transfer and placement of the head frame needs to be completed within the 15minute time frame. The trial's secondary objectives are to determine whether it has any effects on outcomes and quality of life. As part of study participation patients will be asked to complete quality of life questionnaires as well as mini mental status questionnaires. These will be done prior to treatment and at follow up appointments throughout the next 3 years while participating in the study. Patients will be given the option to participate in the optional bio marker blood draw study which would require patients to have blood drawn at three time points, pre-treatment, the day after treatment and at their first follow up visit.

ELIGIBILITY:
Inclusion Criteria

* Metastatic brain tumor referred to radiation oncology for treatment
* Size of the presenting metastatic lesion up to 5.0 cm diameter
* Age > 18 years
* Patients must give informed consent indicating they are aware of the investigational nature of this treatment
* Karnofsky Performance Status > 70% (Zubrod score 0 to 1)
* Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days to start of study therapy
* CBC and CMP within 30 days to start of study therapy
* Chest imaging (Chest Xray or Chest CT) within past 12 months, that does not show any contraindication to hyperbaric therapy (if patient has had any thoracic surgery or other significant event that might have affected the thorax such as trauma, pneumothorax, chest tube insertion, pleurodesis, or thoracentesis and has not had imaging since that event, then the imaging should be repeated).
* Neurosurgery Consult

Exclusion Criteria

* Pregnant women or women of childbearing potential without adequate contraception. Contraception, which can include abstinence, is required since the last menstrual period until completion of SRS.
* Evidence of pneumothorax (Untreated pneumothorax risks tension pneumothorax during ascent in HBO chamber)
* COPD with C02 retention (Such patients can develop respiratory depression as HBO reduces their hypoxemic drive)
* Uncontrolled seizure disorder (Note that patients on adequate antiepileptic medications may receive HBO)
* Claustrophobia resistant to medication (Pre-medication with anxiolytics is generally sufficient for almost all anxious patients undergoing HBO treatment)
* History of middle ear surgery

  * Failure to equalize pressure in the middle ear can cause displacement of middle ear structures with consequent hearing loss
  * To clarify: placement of a tympanostomy tube is not a contraindication to HBO, and in fact may improve tolerability of the procedure
* History of bleomycin administration (HBO can exacerbate interstitial pneumonitis in such patients)
* Current cis-platinum chemotherapy, i.e. therapeutic levels in the bloodstream at the time of HBO therapy. (HBO can increase cytotoxicity of cis-platinum)
* Uncontrolled high blood pressure (HBO can increase systemic vascular resistance)
* Unstable angina or myocardial infarction within the previous 3 months (Increased afterload due to HBO can increase myocardial workload)
* Cardiac EF ≤ 35%

  * Pulmonary edema can arise with HBO in certain patients with severe heart failure
  * In patients with prior history of CHF, subsequent echocardiogram and ECG are required to establish EF>35%
* Treatment with disulfiram (Disulfiram inhibits superoxide dismutase and is not approved for use concomitantly with hyperbaric oxygen therapy)
* Active drug/alcohol dependence or abuse
* Lack of adequate social support structures, e.g. homelessness
* Tumors with potential confounding results on serum marker studies

  * Small cell (neuroendocrine) carcinomas
  * Carcinoid tumors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Hartford, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Hartford AC, Gill GS, Ravi D, Tosteson TD, Li Z, Russo G, Eskey CJ, Jarvis LA, Simmons NE, Evans LT, Williams BB, Gladstone DJ, Roberts DW, Buckey JC Jr. Sensitizing brain metastases to stereotactic radiosurgery using hyperbaric oxygen: A proof-of-principle study. Radiother Oncol. 2022 Dec;177:179-184. doi: 10.1016/j.radonc.2022.10.024. Epub 2022 Oct 28. PMID 36404528

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HBO feasibility subjects were recruited from potential candidates for stereotactic radiosurgery (SRS) treatment at DHMC for brain metastases. Such patients are referred to radiation oncology by practitioners at DHMC and by physicians at outlying hospitals.
  Historic Controls: Retrospective review of previous patients utilizing SRS in the treatment of brain metastases. The control population was selected based on matching variables.
Pre-assignment Details: Adverse events were not collected for historic controls.
Groups:
- HBO Feasibility: Hyperbaric oxygen given at 2.4 ATA for 30 minutes immediately prior to SRS - HBOT for 30 minutes - SRS without prior HBO
- Historic Controls: Retrospective review of previous patients utilizing SRS in the treatment of brain metastases. The matching variables (histology, lesion size, resection status, and calculated GPA) will be used to identify this control population.
Period: Overall Study
Arm/Group | HBO Feasibility | Historic Controls
Started | 22 | 19
HBO Treatment Completed | 19 | 0
Completed (SRS treatment completed) | 19 | 19
Not Completed | 3 | 0
Not completed — Not eligible | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- HBO Feasibility: Hyperbaric oxygen given at 2.4 ATA for 30 minutes immediately prior to SRS - HBOT for 30 minutes - SRS without prior HBO. Demographic information (Race, gender, ethnicity, and age) were collected for only the participants who were prospectively enrolled and provided informed consent.
- Total: Total of all reporting groups
Arm/Group | HBO Feasibility | Historic Controls | Total
Number analyzed (Participants) | 22 | 19 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 10 | 26
  >=65 years | 6 | 9 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 0 | 22
  Unknown or Not Reported | 0 | 19 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 22 | 0 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 19 | 19
Region of Enrollment [Number; unit: participants]
  United States | 22 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: The Average Time From HBO Chamber Exit to SRS beam-on
Description: Time from end of HBO decompression to start of SRS treatment will be measured to determine feasibility. Feasibility is defined as having been achieved if more than 50% of the 20 evaluable patients start SRS treatment within 30 minutes of leaving the HBO tank
Time Frame: Approximately 30 minutes during SRS Treatment Visit
Population: Three (3) participants were screen failures, and did not receive study treatment, and not included in the analysis.
Measure: Mean (Full Range); unit: minutes
Arm/Group | HBO Feasibility
Number analyzed (Participants) | 19
minutes | 8.3 [5 to 12]

2. Secondary Outcome: Overall Survival in Years
Description: Median time to death
Time Frame: 5 year from treatment
Population: Three (3) participants were screen failures, and did not receive study treatment, and not included in the analysis.
Measure: Median (Full Range); unit: Years
Arm/Group | HBO Feasibility | Historic Controls
Number analyzed (Participants) | 19 | 19
Years | 1.42 [0.96 to 2.35] | 1.03 [0.57 to 2.80]

3. Secondary Outcome: Number of Years Until Local Recurrence
Description: Number of years until recurrence of lesion
Time Frame: 5 year from treatment
Population: Three (3) participants were screen failures, and did not receive study treatment, and not included in the analysis.
Measure: Median (Full Range); unit: Years
Arm/Group | HBO Feasibility | Historic Controls
Number analyzed (Participants) | 19 | 19
Years | NA [1.45 to NA] — Insufficient data (only one observed occurrence) | NA [0.70 to NA] — Insufficient data (only one observed occurrence)

4. Secondary Outcome: Number of Years Until Local Recurrence Prior to WBRT
Description: Number of years until local recurrence of lesion prior to whole brain radiation therapy
Time Frame: 5 year from treatment
Population: Three (3) participants were screen failures, and did not receive study treatment, and not included in the analysis.
Measure: Median (Full Range); unit: Years
Arm/Group | HBO Feasibility | Historic Controls
Number analyzed (Participants) | 19 | 19
Years | NA [1.45 to NA] — Insufficient data (only one observed occurrence) | NA [0.70 to NA] — Insufficient data (only one observed occurrence)

5. Secondary Outcome: Number of Participants Developing Intercranial Distant Recurrence
Description: Number of participants who developed intercranial distant recurrence
Time Frame: 5 year from treatment
Population: Three (3) participants were screen failures, and did not receive study treatment, and not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | HBO Feasibility | Historic Controls
Number analyzed (Participants) | 19 | 19
Participants | 9 | 11
Statistical Analysis 1: Comparison: HBO Feasibility vs Historic Controls; Test type: Other; p = 0.76, Kaplan-Meier; Hazard Ratio (HR) = 0.87

6. Secondary Outcome: Number of Months Between SRS Treatment and Whole Brain Radiation Therapy
Time Frame: 5 year from treatment
Population: Three (3) participants were screen failures, and did not receive study treatment, and not included in the analysis. 17 participants in the HBO group, and 14 historical controls did not receive whole brain radiation therapy
Measure: Median (Full Range); unit: Months
Arm/Group | HBO Feasibility | Historic Controls
Number analyzed (Participants) | 2 | 5
Months | 8.5 [1.5 to 23.3] | 5.6 [4.7 to 6.5]

7. Secondary Outcome: Number of Lesions Exhibiting Radionecrosis
Time Frame: 5 year from treatment
Population: Three (3) participants were screen failures, and did not receive study treatment, and not included in the analysis.
Measure: Number; unit: Lesions exhibiting radionecrosis
Units Other Than Participants: Lesions
Arm/Group | HBO Feasibility | Historic Controls
Number analyzed (Participants) | 19 | 19
Number analyzed (Lesions) | 25 | 27
Lesions exhibiting radionecrosis | 5 | 6
Statistical Analysis 1: Comparison: HBO Feasibility vs Historic Controls; Test type: Other; p = 0.76, Kaplan-Meier; Hazard Ratio (HR) = 0.82

8. Other Pre Specified Outcome: Average Score of Quality of Life as Measured by St. Louis University Mental Status Exam (SLUMS) Mental Status Exam (SLUMS)
Description: SLUMS is an 11-item screening tool to evaluate cognitive ability in adults. The SLUMS score ranges from 1-30. For patients with a high school education, the normal range score is 27-30. For mild neurocognitive disorder, the score range is 21-26. Dementia range is 1-20. For patients with less than a high school education the normal range score is 25-30. For mild neurocognitive disorder, the score range is 20-24. Dementia range is 1-19.
  The scores across all time points were averaged to obtain the mean.
Time Frame: Baseline, 4 to 6 weeks after treatment and then every 3 months for a minimum of 1 year, up to 5 years
Population: Three (3) participants were screen failures, and did not receive study treatment, and not included in the analysis. This information was not available for historical controls.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HBO Feasibility
Number analyzed (Participants) | 19
units on a scale | 26.5 (3.4)

9. Other Pre Specified Outcome: Average Score of EORTC Global Health Status (QL2)
Description: Averages score QL2 determined by responses to aggregate combined results of questionnaires (QLQ C-30 and BN-20).
  EORTC Quality of Life Questionnaire C-30 (QLQ C-30): 30-item self-report questionnaire rating items on a 4-point scale (1 "not at all" to 4 "very much") It measures several domains (physical, role, emotional, cognitive, and social functioning, fatigue, pain, nausea and vomiting) and several single items. Scores are averaged for each scale and transformed to 0-100 scale; higher score indicates better QoL on global health status and functional scales and worse QoL on symptom scales and financial difficulty scale.
  EORTC QLQ BN-20 (BN-20): 4 scales comprised of multiple items and 7 single items. All items are rated on a 4-point Likert-type scale, 1=not at all' to 4=very much, and linearly transformed to a 0-100 scale, higher scores indicating more severe symptoms.
  The scores across all time points were averaged to obtain the mean.
Time Frame: Baseline, 4 to 6 weeks after treatment and then every 3 months for a minimum of 1 year, up to 5 years
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- HBO Feasibility: Hyperbaric oxygen given at 2.4 ATA for 30 minutes immediately prior to SRS - HBOT for 30 minutes - SRS without prior HBO. Demographic information (Race, gender, ethnicity, and age) were collected for only the participants who were prospectively enrolled and provided informed consent. Demographic data was not collected for historic controls.
Arm/Group | HBO Feasibility
Number analyzed (Participants) | 19
score on a scale | 66.8 (24.6)

10. Other Pre Specified Outcome: Presence of S100 and NSE (Serum Markers for Tissue Apoptosis and for Neuronal Damage)
Description: Serum markers for tissue apoptosis and for neuronal damage
Time Frame: 24-48 hours after the SRS treatment
Population: Sample donations where optional for the study participants. Insufficient samples were obtained and therefore, samples were not analyzed.
Arm/Group | HBO Feasibility
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AE) for the HBO Feasibility arm will be collected during the period from the initiation of the study procedures until the date of documented death, withdrawal of consent, or the end of the study, whichever occurs first. Collection could span approximately 5 years. Adverse events were not collected for the historic controls.
Description: Symptomatic treatment toxicity: AEs potentially related to intracranial SRS and/or HBO treatments Radiographic evidence for radionecrosis/treatment effects in normal tissue identified by diagnostic radiologist of follow-up MRI imaging. Incidence of WBRT, Incidence of repeat SRS to the index site and a distant site. Local and distant disease recurrence at the treatment site identified by diagnostic radiologist of follow-up MRI imaging. AEs were not collected for historic controls.
Arm/Group | HBO Feasibility | Historic Controls
All-Cause Mortality (participants affected / at risk) | 8/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 5/19 | 6/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HBO Feasibility (N=19) | Historic Controls (N=19)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Cognitive Disturbance (Nervous system disorders) | 1 (1) | 3 (3)
Memory Impairment (Nervous system disorders) | 2 (2) | 2 (2)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Intercranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT01850563/Prot_SAP_000.pdf